CLINICAL TRIAL: NCT04246281
Title: A Randomized, Controlled, Multicenter Trial of Percutaneous Peripheral Nerve Stimulation (PNS) for the Treatment of Back Pain
Brief Title: The RESET Clinical Trial: SPRINT® Peripheral Nerve Stimulation for the Treatment of Back Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SPR Therapeutics, Inc. (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0151-CSP-000; CDMRP-PR170708 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2019-12-19; First posted 2020-01-29 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Low Back Pain; Back Pain
Keywords: Electrical Stimulation; Neuromodulation
MeSH Terms: conditions — Low Back Pain; Back Pain | interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Group 1: Peripheral Nerve Stimulation (PNS) (Active Comparator): Subjects in Group 1 will have leads placed in their lower back. These subjects will then use the SPRINT Peripheral Nerve Stimulation (PNS) System and will receive electrical stimulation for 8 weeks.
  Interventions: Device: SPRINT Peripheral Nerve Stimulation (PNS) System
- Group 2: Standard Interventional Management (Standard of Care) (Active Comparator): Subjects in Group 2 will receive the standard of care. Group 2 subjects may be able to crossover to receive PNS after 12 months from start of treatment (Visit 16).
  Interventions: Procedure: Standard interventional management of low back pain

INTERVENTIONS:
Device: SPRINT Peripheral Nerve Stimulation (PNS) System — The SPRINT System delivers mild electrical stimulation to the nerves in your low back. The SPRINT System includes up to two leads (small wires) that are placed through your skin into your low back. The leads attach to devices worn on your body that deliver stimulation (called Stimulators).
  Arms: Group 1: Peripheral Nerve Stimulation (PNS)
Procedure: Standard interventional management of low back pain — Your doctor will determine which procedure or intervention is appropriate for your back pain. You may receive radiofrequency ablation, spinal cord stimulation, surgery, or another procedure or treatment, as appropriate.
  Arms: Group 2: Standard Interventional Management (Standard of Care)

SUMMARY:
The purpose of this study is to compare standard of care treatments for back pain to electrical stimulation. Stimulation is delivering small amounts of electricity to the nerves in your low back. This study will use a device called the SPRINT Peripheral Nerve Stimulation (PNS) System. The device is cleared by the FDA for up to 60 days of use for the relief of chronic or acute pain (including back pain)

ELIGIBILITY:
Key Inclusion Criteria:

* Chronic low back pain

Key Exclusion Criteria:

* Body Mass Index (BMI) > 40
* Prior lumbar surgery
* Implanted electronic device
* Pregnant

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2020-06-17 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Reduction in average pain intensity | Up to 3-months after Start of Therapy (SOT)
  Average pain is measured using question 5 from the Brief Pain Inventory- Short Form (BPI-5). BPI-5 is a scale of 0 to 10 where 0 represents no pain and 10 represents worst pain.
Study-Related Adverse Events (AEs) | During the Medial Branch Block procedure
  Occurrence and type of study-related AEs
Study-Related Adverse Events (AEs) | During the Lead Placement procedure (SOT)
  Occurrence and type of study-related AEs
Study-Related Adverse Events (AEs) | 1-week post-SOT
  Occurrence and type of study-related AEs
Study-Related Adverse Events (AEs) | 2-weeks post-SOT
  Occurrence and type of study-related AEs
Study-Related Adverse Events (AEs) | 3-weeks post-SOT
  Occurrence and type of study-related AEs
Study-Related Adverse Events (AEs) | 4-weeks post-SOT
  Occurrence and type of study-related AEs
Study-Related Adverse Events (AEs) | 5-weeks post-SOT
  Occurrence and type of study-related AEs
Study-Related Adverse Events (AEs) | 6-weeks post-SOT
  Occurrence and type of study-related AEs
Study-Related Adverse Events (AEs) | 7-weeks post-SOT
  Occurrence and type of study-related AEs
Study-Related Adverse Events (AEs) | 8-weeks post-SOT
  Occurrence and type of study-related AEs
Study-Related Adverse Events (AEs) | 3-months post-SOT
  Occurrence and type of study-related AEs
Study-Related Adverse Events (AEs) | 6-months post-SOT
  Occurrence and type of study-related AEs
Study-Related Adverse Events (AEs) | 9-months post-SOT
  Occurrence and type of study-related AEs
Study-Related Adverse Events (AEs) | 12-months post-SOT
  Occurrence and type of study-related AEs
Study-Related Adverse Events (AEs) | 18-months post-SOT
  Occurrence and type of study-related AEs
Study-Related Adverse Events (AEs) | 24-months post-SOT
  Occurrence and type of study-related AEs

SECONDARY OUTCOMES:
Reduction in pain interference | Baseline, 3-months after SOT
  Measured using question 9 from the Brief Pain Inventory- Short Form. This question asks the subject to rate the degree to which their pain has interfered with general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life on a scale of 0 to 10, where 0 is "does not interfere" and 10 is "completely interferes" within the last week.
Reduction in disability | Baseline, 3-months after SOT
  Measured using the Oswestry Disability Index (ODI). The ODI asks subjects to rate how their back pain impacts ten components of everyday life. For each section, the answers correlate to a scale which ranges from 0 to 5, where 0 is no disability and 5 is maximum disability.
Durability of reductions in pain intensity | Baseline, 6-months after SOT, 9-months after SOT, 12-months after SOT, 18-months after SOT, 24 months after SOT
  Measured using question 5 from the Brief Pain Inventory- Short Form (BPI-5). BPI-5 is a scale of 0 to 10 where 0 represents no pain and 10 represents worst pain.
Reduction in worst pain intensity | Baseline, 3-months after SOT
  Measured using question 3 from the Brief Pain Inventory- Short Form (BPI-3). BPI-3 is a scale of 0 to 10 where 0 represents no pain and 10 represents worst pain.
Patient Global Impression of Change | 3-months after SOT
  Measured using the Patient Global Impression of Change (PGIC) survey. The PGIC scale asks subjects to rate their improvement with treatment on a 7-point scale (centered at 4) that ranges from "very much worse" to "very much improved" relative to baseline.
Change in health-related quality of life | Baseline, 3-months after SOT
  Measured using the EQ-5D survey. The EQ-5D is a five-level scale. Each level is coded from 1 to 5, where 1 indicates no problems and 5 indicates extreme problems. The EQ-5D also includes a 0 to 100 scale for health status, where 0 indicates "the worst health you can imagine" and 100 indicates "the best health you can imagine".
Change in analgesic medication usage | Baseline, 3-months after SOT
  Analgesic medication consumption will be collected.

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - IPM Medical Group, Walnut Creek, California
  - Denver Back Pain Specialists, Greenwood Village, Colorado
  - International Spine, Pain & Performance Center, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia
  - Northwest Speciality Hospital, Post Falls, Idaho
  - Millennium Pain Center, Bloomington, Illinois
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Premier Pain Centers, Shrewsbury, New Jersey
  - Duke University, Durham, North Carolina
  - Center for Clinical Research, Winston-Salem, North Carolina
  - The Ohio State University, Columbus, Ohio
  - Main Line Spine, King of Prussia, Pennsylvania
  - Institute of Precision Pain Medicine, Corpus Christi, Texas
  - University of Utah, Salt Lake City, Utah
  - Virginia iSpine Physicians, Richmond, Virginia
  - Hunter Holmes McGuire Veterans Affairs Medical Center, Richmond, Virginia
  - Spine and Nerve Center of St. Francis Hospital, Charleston, West Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor's Website — http://www.sprintpns.com

DOCUMENTS (1):
  • Study Protocol (2024-04-04): https://cdn.clinicaltrials.gov/large-docs/81/NCT04246281/Prot_000.pdf